CLINICAL TRIAL: NCT00822523
Title: Strain Gauge Feasibility Assessment & Correlation With Compound Muscle Action Potential & Surface Electromyogram Parameters Before & After a Single Intramuscular Injection of Botulinum Toxin Type A Into Extensor Digitorum Brevis Muscle
Brief Title: Assessment of the Effect of Botulinum Toxin in Extensor Digitorum Brevis Via Strain Gauge and Nerve Conduction Studies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Loma Linda University (Other)
Collaborators: Allergan (Industry)
Responsible Party: Principal Investigator, Gordon Peterson, MD, Loma Linda University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: 58360
Record Dates: First submitted 2009-01-12; First posted 2009-01-14 (Estimated); Results first posted 2016-08-31 (Estimated); Last update posted 2018-09-05 (Actual); Status verified 2018-08

CONDITIONS: Muscle Strength; Botulinum Toxins, Type A
MeSH Terms: interventions — Botulinum Toxins, Type A; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Botulinum toxin type A, 20 units (Experimental): Single intramuscular (into extensor digitorum brevis muscle of the foot) dose of Botulinum toxin type A, 20 units
  Interventions: Drug: Botulinum Toxin, Type A
- Botulinum toxin, type A, 2 units (Experimental): Single intramuscular (into extensor digitorum brevis muscle of the foot) dose of Botulinum toxin type A, 2 units
  Interventions: Drug: Botulinum Toxin, Type A
- Placebo (Placebo Comparator): Saline, Single dose, Intramuscular injection into right EDB
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Botulinum Toxin, Type A — 20 units, single dose, intramuscular in right EDB muscle
  Other Names: BOTOX
  Arms: Botulinum toxin type A, 20 units
Drug: Botulinum Toxin, Type A — 2 units, single dose, intramuscular to right EDB muscle
  Other Names: BOTOX
  Arms: Botulinum toxin, type A, 2 units
Drug: Saline — Single Dose, Intramuscular into right EDB muscle
  Other Names: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this feasibility study is to determine if temporary weakness of a small foot muscle caused by local injection of botulinum toxin into that muscle can be measured with a strain gauge in addition to the previously known valid measurements via nerve conduction studies and surface electromyogram.

DETAILED DESCRIPTION:
Purpose/Hypothesis:

Verify the validity and reliability of strain gauge assessment of strength of extensor digitorum brevis (EDB) muscle compared to compound muscle action potential (CMAP) size from EDB and surface electromyography (SEMG) data from EDB after injection of botulinum toxin into EDB

1. Primary Outcome Measure:

   Change in measured strength (using strain gauges) of dorsiflexion of digits 3 and 4 ("strength of EDB") after vs. before botulinum toxin injection into EDB
2. Secondary Outcome Measures:

   1. Change in CMAP (with standard reference electrode location and with an "inactive" reference electrode location) from EDB after vs. before botulinum toxin injection into EDB;
   2. Change in SEMG parameters from EDB, tibialis anterior (TA), and extensor digitorum longus (EDL) after vs. before botulinum toxin injection into EDB

STUDY DESIGN:

1. Overview:

   Single intramuscular injection of botulinum toxin or placebo (placebo or BOTOX 2 units or BOTOX 20 units, each with a total volume of 0.1 ml) intramuscular into right EDB on Day 0. Strain gauge data and SEMG data from TA and EDL are obtained at each evaluation time: Baseline (3 separate times prior to Day 0 after at least 5 separate training sessions for the strain gauges); Day 1; Day 2; Day 4 (during anticipated rapid change); Day 14 (+/-1 day) (at clinical nadir); Day 21 (+/-1 day) (another day at clinical nadir); and Month 4 (when clinical recovery from the effect of BOTOX should have occurred); CMAP & SEMG data from EDB are obtained at Baseline; Day 4 (close to nadir of CAMP); Day 14 (at nadir of CAMP) and/or Day 21 (at nadir of CAMP); and Month 4 (when clinical recovery from the effect of BOTOX should have occurred but CMAP should not have recovered).
2. Protocol:

Single-center, Double-Blind, Randomized, Pilot Trial Total Sample Size: 12-15

Treatment Groups:

BOTOX Single Dose 20 units IM in EDB in 0.1 ml BOTOX Single Dose 2 units IM in EDB in 0.1 ml Placebo (Saline) Single Dose IM in EDB in 0.1 ml

Estimated Time to Enroll:

0-3 months

Estimated Study Duration:

4-6 months

ELIGIBILITY:
Inclusion Criteria:

* Normal, healthy, male or female subjects, 18 to 54 years of age.
* Written informed consent has been obtained.
* Females with child-bearing potential have a negative urine pregnancy test and agree to use a reliable form of contraception during the study.
* Ability to follow study instructions and likely to complete all required visits.
* Written authorization for Use and Release of Health and Research Study Information has been obtained.

Exclusion Criteria:

* Abnormality by focused history and examination including the presence of foot deformity.
* Abnormal (as determined by the investigator) screening nerve conduction studies of the lower limbs.
* Identification of anomalous innervation of right EDB via screening nerve conduction studies.
* The subject having a foot which does not adequately fit in the modified ankle-foot orthosis used with the strain gauge.
* The subject having a foot in which anatomic bone landmarks cannot be adequately identified.
* Body mass index (BMI) greater than 30.
* History of significant (as determined by the investigator) lower limb injury or lower limb surgery
* Any uncontrolled clinically significant medical condition.
* Known allergy or sensitivity to any of the components in the study medication.
* Females with a positive pregnancy test, or who are breast-feeding, planning a pregnancy during the study, who think that they may be pregnant at the start of the study, or females of childbearing potential who are unable or unwilling to use a reliable form of contraception during the study.
* Concurrent participation in another investigational drug or device study or participation within 3 months prior to study.
* Treatment with botulinum toxin of any serotype prior to enrollment in study or prior clinical botulism.
* Any medical condition that may put the subject at increased risk with exposure to BOTOX including diagnosed myasthenia gravis, Lambert-Eaton myasthenic syndrome, amyotrophic lateral sclerosis, or any other disorder that might interfere with neuromuscular function.
* Evidence of alcohol abuse, drug abuse, or other relevant neuropsychiatric condition.
* Infection or skin disorder at an anticipated injection site.
* Any condition or situation that, in the investigator's opinion, may put the subject at significant risk, confound the study results (e.g. variable strength on serial testing during screening examination; or foot, toe, or ankle pain that may limit full participation in muscle strength testing), or interfere significantly with the subject's participation in the study.

Ages: 18 Years to 54 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2009-01; Primary Completion 2009-03 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gordon W Peterson, MD, Principal Investigator — Loma Linda University
Locations (2):
- United States (2):
  - Electromyography Laboratory, Loma Linda University Medical Center, Loma Linda, California
  - Loma Linda University, Loma Linda, California

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sloop RR, Escutin RO, Matus JA, Cole BA, Peterson GW. Dose-response curve of human extensor digitorum brevis muscle function to intramuscularly injected botulinum toxin type A. Neurology. 1996 May;46(5):1382-6. doi: 10.1212/wnl.46.5.1382. PMID 8628486
- [Background] Hamjian JA, Walker FO. Serial neurophysiological studies of intramuscular botulinum-A toxin in humans. Muscle Nerve. 1994 Dec;17(12):1385-92. doi: 10.1002/mus.880171207. PMID 7969239

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Botulinum Toxin Type A, 20 Units | Botulinum Toxin, Type A, 2 Units | Placebo
Started | 5 | 4 | 4
Completed | 5 | 4 | 4
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Botulinum Toxin Type A, 20 Units | Botulinum Toxin, Type A, 2 Units | Placebo | Total
Number analyzed (Participants) | 5 | 4 | 4 | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 5 | 4 | 4 | 13
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 31 (5.9) | 26.8 (2.1) | 29.5 (2.0) | 29.2 (2.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 1 | 5
  Male | 3 | 2 | 3 | 8
Region of Enrollment [Number; unit: participants]
  United States | 5 | 4 | 4 | 13

OUTCOME MEASURES:

1. Primary Outcome: Change in Measured Force (Change From Baseline) (Using Strain Gauges) of Dorsiflexion of Digits 2 and 3 ("Force of EDB") After vs. Before Botulinum Toxin Injection Into EDB
Description: The force of dorsiflexion of the combination of digits 2 and 3 (at the same time using a single loop) of the foot were measured using a strain gauge after and before the administration of Botulinum Neurotoxin type A (BoNT/A) or placebo. The baseline value was the mean of the 3 values for force obtained prior to injection of BoNT/A. The baseline was compared with the subsequent values.
Time Frame: Baseline (3 times) then following single injection of botulinum toxin into EDB with testing at Day 1, Day 2, Day 4, Day 14, Day 21, and Month 4
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Botulinum Toxin Type A, 20 Units | Botulinum Toxin, Type A, 2 Units | Placebo
Number analyzed (Participants) | 5 | 4 | 4
kg
  Baseline | 7.63 (3.31) | 5.16 (1.48) | 10.43 (5.33)
  Day 1 | 7.85 (3.76) | 4.28 (1.02) | 12.22 (8.26)
  Day 2 | 9.37 (3.21) | 4.46 (1.22) | 10.88 (7.21)
  Day 4 | 10.42 (6.56) | 4.85 (0.75) | 11.38 (9.59)
  Day 14 | 7.89 (3.7) | 4.75 (1.00) | 13.46 (8.49)
  Day 21 | 9.60 (4.51) | 4.20 (2.11) | 11.88 (6.82)
  Month 4 | 7.62 (4.44) | 5.27 (1.37) | 11.23 (6.92)
Statistical Analysis 1: Comparison: Botulinum Toxin Type A, 20 Units vs Botulinum Toxin, Type A, 2 Units vs Placebo; Two sample t-test comparing baseline and day 1 H0: There is no change in mean force between baseline and day 1 HA: There is change in mean force between baseline and day 1; Test type: Superiority or Other; p = 0.61, t-test, 2 sided
Statistical Analysis 2: Comparison: Botulinum Toxin Type A, 20 Units vs Botulinum Toxin, Type A, 2 Units vs Placebo; Two sample t-test comparing baseline and day 2 H0: There is no change in mean force between baseline and day 2 HA: There is change in mean force between baseline and day 2; Test type: Superiority or Other; p = 0.787, t-test, 2 sided
Statistical Analysis 3: Comparison: Botulinum Toxin Type A, 20 Units vs Botulinum Toxin, Type A, 2 Units vs Placebo; Two sample t-test comparing baseline and day 4 H0: There is no change in mean force between baseline and day 4 HA: There is change in mean force between baseline and day 4; Test type: Superiority or Other; p = 0.234, t-test, 2 sided
Statistical Analysis 4: Comparison: Botulinum Toxin Type A, 20 Units vs Botulinum Toxin, Type A, 2 Units vs Placebo; Two sample t-test comparing baseline and day 14 H0: There is no change in mean force between baseline and day 14 HA: There is change in mean force between baseline and day 14; Test type: Superiority or Other; p = 0.256, t-test, 2 sided
Statistical Analysis 5: Comparison: Botulinum Toxin Type A, 20 Units vs Botulinum Toxin, Type A, 2 Units vs Placebo; Two sample t-test comparing baseline and day 21 H0: There is no change in mean force between baseline and day 21 HA: There is change in mean force between baseline and day 21; Test type: Superiority or Other; p = 0.292, t-test, 2 sided
Statistical Analysis 6: Comparison: Botulinum Toxin Type A, 20 Units vs Botulinum Toxin, Type A, 2 Units vs Placebo; Two sample t-test comparing baseline and month 4 H0: There is no change in mean force between baseline and month 4 HA: There is change in mean force between baseline and month 4; Test type: Superiority or Other; p = 0.589, t-test, 2 sided

2. Secondary Outcome: Stability of Baseline Measurements of Force
Description: The force of dorsiflexion of the combination of digits 2 and 3 (at the same time using a single loop) of the foot were measured using a strain gauge on three different days prior to injection of BoNT/A or placebo. On each of the three days of baseline testing, the force was defined as the mean of three different measurements, separated by at least 1 minute from another measurement.
Time Frame: Baseline 1 (mean of 3 measurement on the same day of testing) compared with Baseline 2 (mean of 3 measurement on the same day of testing) on a second day compared with Baseline 3 (mean of 3 measurement on the same day of testing)
Population: Normal controls at baseline before BoNT/A injected
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Botulinum Toxin Type A, 20 Units | Botulinum Toxin, Type A, 2 Units | Placebo
Number analyzed (Participants) | 5 | 4 | 4
kg
  Baseline 1 | 7.78 (4.29) | 4.83 (1.21) | 11.15 (5.28)
  Baseline 2 | 7.58 (3.38) | 5.28 (1.81) | 9.82 (5.29)
  Baseline 3 | 7.51 (2.47) | 5.35 (1.70) | 10.32 (5.46)
Statistical Analysis 1: Comparison: Botulinum Toxin Type A, 20 Units vs Botulinum Toxin, Type A, 2 Units vs Placebo; Repeated measure ANOVA assessing change in the three baseline force measurements H0: There no significant difference in the three baseline force measurements HA: There is a significant difference in the three baseline force measurements; Test type: Superiority or Other; p = 0.636, Repeated measure ANOVA
Statistical Analysis 2: Comparison: Botulinum Toxin Type A, 20 Units vs Botulinum Toxin, Type A, 2 Units vs Placebo; Repeated measure ANOVA assessing change in baseline force by treatment arm. H0: There is no difference in mean baseline force by treatment arm HA: There is a difference in mean baseline force by treatment arm; Test type: Superiority or Other; p = 0.178, Repeated measure ANOVA

3. Secondary Outcome: Difference in Force From Day 14 to Day 21
Description: The force of dorsiflexion of the combination of digits 2 and 3 (at the same time using a single loop) of the foot were measured using a strain gauge after and before the administration of Botulinum Neurotoxin type A (BoNT/A). The force at each day of testing was the mean of the 3 values for force obtained on that day. Value is percent change from baseline. Comparison is made between the percent change from baseline force and the force on Day 14 in each group vs. the percent change from baseline force and the force on Day 21 in each group.
Time Frame: Force measured at Day 14 after BoNT/A injction into EDB and Force measured at Day 21 after BoNT/A injction into EDB.
Measure: Mean (Standard Deviation); unit: percent change from baseline
Arm/Group | Botulinum Toxin Type A, 20 Units | Botulinum Toxin, Type A, 2 Units | Placebo
Number analyzed (Participants) | 5 | 4 | 4
percent change from baseline
  Day 14 | 4.57 (19.66) | -4.81 (20.94) | 22.66 (32.22)
  Day 21 | 27.01 (27.44) | -19.58 (41.04) | 15.15 (32.15)
Statistical Analysis 1: Comparison: Botulinum Toxin Type A, 20 Units vs Botulinum Toxin, Type A, 2 Units vs Placebo; Repeated measure ANOVA assessing percent change (from baseline) in force for contrast of day 14 and day 21 H0: There is no difference in percent change in force between day 14 and day 21 HA: There is a difference in percent change in force between day 14 and day 21; Test type: Superiority or Other; p = 0.995, Repeated measure ANOVA
Statistical Analysis 2: Comparison: Botulinum Toxin Type A, 20 Units vs Botulinum Toxin, Type A, 2 Units vs Placebo; Repeated measure ANOVA assessing percent change in force from baseline for day 14 and 21 by treatment arm. H0: There is no significant different in percent change in force by treatment arm HA: There is a significant different in percent change in force by treatment arm; Test type: Superiority or Other; p = 0.2088, Repeated measure ANOVA

4. Secondary Outcome: Number of Participants With Serious Adverse Effects to onabotulinumtoxinA (Botulinum Type A Neurotoxin)
Time Frame: At each visit for nerve conduction studies following injection of onabotulinumtoxinA (botulinum type A neurotoxin) into EDB (Day 0; Day 4; Day 14; Month 4)
Measure: Number; unit: participants
Arm/Group | Botulinum Toxin Type A, 20 Units | Botulinum Toxin, Type A, 2 Units | Placebo
Number analyzed (Participants) | 5 | 4 | 4
participants | 0 | 0 | 0

5. Secondary Outcome: Correlation in Percent Change of the CMAP (With Standard Reference Electrode Location) From EDB After vs. Before Botulinum Toxin Injection Into EDB vs. Percent Change Surface Electromyography (as Measured by Root Mean Squared With 1000 ms Window).
Description: Measure the percent change of the Compound Muscle Action Potential (CMAP) Amplitude from extensor digitorum brevis (EDB) with the reference electrode in the standard location at the base of the ipsilateral 5th toe after injection of BoNT/A into EDB compared with before injection of BoNT/A. Each CMAP represents the mean of 3 individual measurements of the CMAP at that timepoint. In order to facilitate comparison from one subject to the next, the CMAP is then converted into percent change from baseline for that subject. CMAP percent change is then correlated with the percent change in the Surface Electromyography as measured by the Root Mean Squared with 1000 millisecond window at the same time points after injection. Group with injection of 20 units BoNT/A is used.
Time Frame: Mean of 3 measurements on the same day of testing following single injection of botulinum toxin into EDB with testing at Day 4; Day 14; and Month 4 each compared with Baseline measurement
Population: Analysis of the 2 Units Botox and placebo arms was to be done only if the arm with 20 Units Botox showed significant changes in the strain gauge measurements.
Measure: Mean (Standard Deviation); unit: percent change from baseline
Groups:
- CMAP (Standard) With Botulinum Toxin Type A, 20 Units: Compound muscle action potential (CMAP) with reference electrode in the standard location at the base of the ipsilateral 5th toe
  Single intramuscular (into extensor digitorum brevis muscle of the foot) dose of Botulinum toxin type A, 20 units
  Botulinum Toxin, Type A: 20 units, single dose, intramuscular in right EDB muscle
- Surface EMG RMS-1000 With Botulinum Toxin Type A, 20 Units: Surface Electromyography (Surface EMG) measured as the RMS (Root Mean Squared) with 1000 ms interval
  Single intramuscular (into extensor digitorum brevis muscle of the foot) dose of Botulinum toxin type A, 20 units
  Botulinum Toxin, Type A: 20 units, single dose, intramuscular in right EDB muscle
Arm/Group | CMAP (Standard) With Botulinum Toxin Type A, 20 Units | Surface EMG RMS-1000 With Botulinum Toxin Type A, 20 Units
Number analyzed (Participants) | 5 | 5
percent change from baseline
  Day 4 | -53.81 (21.81) | -42.43 (19.82)
  Day 14 | -63.78 (21.77) | -52.35 (27.17)
  Month 4 | -48.38 (26.16) | -39.76 (11.26)
Statistical Analysis 1: Comparison: CMAP (Standard) With Botulinum Toxin Type A, 20 Units vs Surface EMG RMS-1000 With Botulinum Toxin Type A, 20 Units; Day 4; Test type: Superiority or Other; p = 0.0374, Spearman Correlation Test; r value = 0.9
Statistical Analysis 2: Comparison: CMAP (Standard) With Botulinum Toxin Type A, 20 Units vs Surface EMG RMS-1000 With Botulinum Toxin Type A, 20 Units; Day 14; Test type: Superiority or Other; p = 0.188, Spearman Correlation Test; r value = 0.7
Statistical Analysis 3: Comparison: CMAP (Standard) With Botulinum Toxin Type A, 20 Units vs Surface EMG RMS-1000 With Botulinum Toxin Type A, 20 Units; Month 4; Test type: Superiority or Other; p = 0.104, Spearman Correlation Test; r value = 0.8

6. Secondary Outcome: Percent Change of the Surface Electromyogram (SEMG) MRV-500 From EDB After vs. Before Botulinum Toxin Injection Into EDB.
Description: Measure the percent change of the Surface Electromyogram (SEMG) as measured by the Mean Rectified Voltage (MRV) with a window of 500 ms from extensor digitorum brevis (EDB) with the reference electrode in the standard location at the base of the ipsilateral 5th toe after injection of BoNT/A into EDB compared with before injection of BoNT/A or placebo. Each MRV represents the mean of 3 individual measurements of the MRV at that timepoint with measurements at least 60 seconds apart. In order to facilitate comparison from one subject to the next, the MRV is then converted into percent change from baseline for that subject.
Time Frame: Baseline (mean of 3 measurement on the same day of testing) then following single injection of botulinum toxin into EDB with testing at Day 4; Day 14; and Month 4
Measure: Mean (Standard Deviation); unit: percent change from baseline
Arm/Group | Botulinum Toxin Type A, 20 Units | Botulinum Toxin, Type A, 2 Units | Placebo
Number analyzed (Participants) | 5 | 4 | 4
percent change from baseline
  Day 4 | -40.4 (20.0) | -44.4 (7.6) | -4.1 (69.6)
  Day 14 | -50.8 (27.4) | -52.2 (14.6) | 0.7 (38.2)
  Month 4 | -39.2 (9.4) | -19.8 (25.0) | -28.6 (56.4)

7. Secondary Outcome: Correlation in Percent Change of the CMAP (With Standard Reference Electrode Location) From EDB After vs. Before Botulinum Toxin Injection Into EDB vs. Percent Change Surface Electromyography (as Measured by Root Mean Squared With 500 ms Window).
Description: Measure the percent change of the Compound Muscle Action Potential (CMAP) Amplitude from extensor digitorum brevis (EDB) with the reference electrode in the standard location at the base of the ipsilateral 5th toe after injection of BoNT/A into EDB compared with before injection of BoNT/A. Each CMAP represents the mean of 3 individual measurements of the CMAP at that timepoint. In order to facilitate comparison from one subject to the next, the CMAP is then converted into percent change from baseline for that subject. CMAP percent change is then correlated with the percent change in the Surface Electromyography as measured by the Root Mean Squared with 500 millisecond window at the same time points after injection. Group with injection of 20 units BoNT/A is used.
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: percent change from baseline
Groups:
- Surface EMG RMS-500 With Botulinum Toxin Type A, 20 Units: Surface Electromyography (Surface EMG) measured as the RMS (Root Mean Squared) with 500 ms interval
  Single intramuscular (into extensor digitorum brevis muscle of the foot) dose of Botulinum toxin type A, 20 units
  Botulinum Toxin, Type A: 20 units, single dose, intramuscular in right EDB muscle
Arm/Group | CMAP (Standard) With Botulinum Toxin Type A, 20 Units | Surface EMG RMS-500 With Botulinum Toxin Type A, 20 Units
Number analyzed (Participants) | 5 | 5
percent change from baseline
  Day 4 | -53.81 (21.81) | -42.09 (21.19)
  Day 14 | -63.78 (21.77) | -51.94 (28.01)
  Month 4 | -48.38 (26.16) | -40.67 (11.48)
Statistical Analysis 1: Comparison: CMAP (Standard) With Botulinum Toxin Type A, 20 Units vs Surface EMG RMS-500 With Botulinum Toxin Type A, 20 Units; Day 4; Test type: Superiority or Other; p = 0.0374, Spearman Correlation Test; r value = 0.9
Statistical Analysis 2: Comparison: CMAP (Standard) With Botulinum Toxin Type A, 20 Units vs Surface EMG RMS-500 With Botulinum Toxin Type A, 20 Units; Day 14; Test type: Superiority or Other; p = 0.188, Spearman Correlation Test; r value = 0.7
Statistical Analysis 3: Comparison: CMAP (Standard) With Botulinum Toxin Type A, 20 Units vs Surface EMG RMS-500 With Botulinum Toxin Type A, 20 Units; Month 4; Test type: Superiority or Other; p = 0.0374, Spearman Correlation Test; r value = 0.9

8. Secondary Outcome: Correlation in Percent Change of the CMAP (With Standard Reference Electrode Location) From EDB After vs. Before Botulinum Toxin Injection Into EDB vs. Percent Change Surface Electromyography (as Measured by Root Mean Squared With 200 ms Window).
Description: Measure the percent change of the Compound Muscle Action Potential (CMAP) Amplitude from extensor digitorum brevis (EDB) with the reference electrode in the standard location at the base of the ipsilateral 5th toe after injection of BoNT/A into EDB compared with before injection of BoNT/A. Each CMAP represents the mean of 3 individual measurements of the CMAP at that timepoint. In order to facilitate comparison from one subject to the next, the CMAP is then converted into percent change from baseline for that subject. CMAP percent change is then correlated with the percent change in the Surface Electromyography as measured by the Root Mean Squared with 200 millisecond window at the same time points after injection. Group with injection of 20 units BoNT/A is used.
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: percent change from baseline
Groups:
- Surface EMG RMS-200 With Botulinum Toxin Type A, 20 Units: Surface Electromyography (Surface EMG) measured as the RMS (Root Mean Squared) with 200 ms interval
  Single intramuscular (into extensor digitorum brevis muscle of the foot) dose of Botulinum toxin type A, 20 units
  Botulinum Toxin, Type A: 20 units, single dose, intramuscular in right EDB muscle
Arm/Group | CMAP (Standard) With Botulinum Toxin Type A, 20 Units | Surface EMG RMS-200 With Botulinum Toxin Type A, 20 Units
Number analyzed (Participants) | 5 | 5
percent change from baseline
  Day 4 | -53.81 (21.81) | -39.89 (22.65)
  Day 14 | -63.78 (21.77) | -51.75 (28.52)
  Month 4 | -48.38 (26.16) | -39.90 (12.43)
Statistical Analysis 1: Comparison: CMAP (Standard) With Botulinum Toxin Type A, 20 Units vs Surface EMG RMS-200 With Botulinum Toxin Type A, 20 Units; Day 4; Test type: Superiority or Other; p = 0.0374, Spearman Correlation Test; r value = 0.9
Statistical Analysis 2: Comparison: CMAP (Standard) With Botulinum Toxin Type A, 20 Units vs Surface EMG RMS-200 With Botulinum Toxin Type A, 20 Units; Day 14; Test type: Superiority or Other; p = 0.188, Spearman Correlation Test; r value = 0.7
Statistical Analysis 3: Comparison: CMAP (Standard) With Botulinum Toxin Type A, 20 Units vs Surface EMG RMS-200 With Botulinum Toxin Type A, 20 Units; Month 4; Test type: Superiority or Other; p = 0.188, Spearman Correlation Test; r value = 0.7

9. Secondary Outcome: Correlation in Percent Change of the CMAP (With Standard Reference Electrode Location) From EDB After vs. Before Botulinum Toxin Injection Into EDB vs. Percent Change Surface Electromyography (as Measured by Mean Rectified Voltage With 1000 ms Window).
Description: Measure the percent change of the Compound Muscle Action Potential (CMAP) Amplitude from extensor digitorum brevis (EDB) with the reference electrode in the standard location at the base of the ipsilateral 5th toe after injection of BoNT/A into EDB compared with before injection of BoNT/A. Each CMAP represents the mean of 3 individual measurements of the CMAP at that timepoint. In order to facilitate comparison from one subject to the next, the CMAP is then converted into percent change from baseline for that subject. CMAP percent change is then correlated with the percent change in the Surface Electromyography as measured by the Mean Rectified Voltage with 1000 millisecond window at the same time points after injection. Group with injection of 20 units BoNT/A is used.
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: percent change from baseline
Groups:
- Surface EMG MRV-1000 With Botulinum Toxin Type A, 20 Units: Surface Electromyography (Surface EMG) measured as the MRV (Mean Rectified Voltage) with 1000 ms interval
  Single intramuscular (into extensor digitorum brevis muscle of the foot) dose of Botulinum toxin type A, 20 units
  Botulinum Toxin, Type A: 20 units, single dose, intramuscular in right EDB muscle
Arm/Group | CMAP (Standard) With Botulinum Toxin Type A, 20 Units | Surface EMG MRV-1000 With Botulinum Toxin Type A, 20 Units
Number analyzed (Participants) | 5 | 5
percent change from baseline
  Day 4 | -53.81 (21.81) | -40.92 (18.90)
  Day 14 | -63.78 (21.77) | -51.03 (26.56)
  Month 4 | -48.38 (26.16) | -37.86 (9.45)
Statistical Analysis 1: Comparison: CMAP (Standard) With Botulinum Toxin Type A, 20 Units vs Surface EMG MRV-1000 With Botulinum Toxin Type A, 20 Units; Day 4; Test type: Superiority or Other; p = 0.0374, Spearman Correlation Test; r value = 0.9
Statistical Analysis 2: Comparison: CMAP (Standard) With Botulinum Toxin Type A, 20 Units vs Surface EMG MRV-1000 With Botulinum Toxin Type A, 20 Units; Day 14; Test type: Superiority or Other; p = 0.188, Spearman Correlation Test; r value = 0.7
Statistical Analysis 3: Comparison: CMAP (Standard) With Botulinum Toxin Type A, 20 Units vs Surface EMG MRV-1000 With Botulinum Toxin Type A, 20 Units; Month 4; Test type: Superiority or Other; p = 0.391, Spearman Correlation Test; r value = 0.5

10. Secondary Outcome: Correlation in Percent Change of the CMAP (With Standard Reference Electrode Location) From EDB After vs. Before Botulinum Toxin Injection Into EDB vs. Percent Change Surface Electromyography (as Measured by Mean Rectified Voltage With 500 ms Window).
Description: Measure the percent change of the Compound Muscle Action Potential (CMAP) Amplitude from extensor digitorum brevis (EDB) with the reference electrode in the standard location at the base of the ipsilateral 5th toe after injection of BoNT/A into EDB compared with before injection of BoNT/A. Each CMAP represents the mean of 3 individual measurements of the CMAP at that timepoint. In order to facilitate comparison from one subject to the next, the CMAP is then converted into percent change from baseline for that subject. CMAP percent change is then correlated with the percent change in the Surface Electromyography as measured by the Mean Rectified Voltage with 500 millisecond window at the same time points after injection. Group with injection of 20 units BoNT/A is used.
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: percent change from baseline
Groups:
- Surface EMG MRV-500 With Botulinum Toxin Type A, 20 Units: Surface Electromyography (Surface EMG) measured as the MRV (Mean Rectified Voltage) with 500 ms interval
  Single intramuscular (into extensor digitorum brevis muscle of the foot) dose of Botulinum toxin type A, 20 units
  Botulinum Toxin, Type A: 20 units, single dose, intramuscular in right EDB muscle
Arm/Group | CMAP (Standard) With Botulinum Toxin Type A, 20 Units | Surface EMG MRV-500 With Botulinum Toxin Type A, 20 Units
Number analyzed (Participants) | 5 | 5
percent change from baseline
  Day 4 | -53.81 (21.81) | -40.44 (20.00)
  Day 14 | -63.78 (21.77) | -50.72 (27.40)
  Month 4 | -48.38 (26.16) | -39.22 (9.42)
Statistical Analysis 1: Comparison: CMAP (Standard) With Botulinum Toxin Type A, 20 Units vs Surface EMG MRV-500 With Botulinum Toxin Type A, 20 Units; Day 4; Test type: Superiority or Other; p = 0.0374, Spearman Correlation Test; r value = 0.9
Statistical Analysis 2: Comparison: CMAP (Standard) With Botulinum Toxin Type A, 20 Units vs Surface EMG MRV-500 With Botulinum Toxin Type A, 20 Units; Day 14; Test type: Superiority or Other; p = 0.188, Spearman Correlation Test; r value = 0.7
Statistical Analysis 3: Comparison: CMAP (Standard) With Botulinum Toxin Type A, 20 Units vs Surface EMG MRV-500 With Botulinum Toxin Type A, 20 Units; Month 4; Test type: Superiority or Other; p = 0.0374, Spearman Correlation Test; r value = 0.9

11. Secondary Outcome: Correlation in Percent Change of the CMAP (With Standard Reference Electrode Location) From EDB After vs. Before Botulinum Toxin Injection Into EDB vs. Percent Change Surface Electromyography (as Measured by Mean Rectified Voltage With 200 ms Window).
Description: Measure the percent change of the Compound Muscle Action Potential (CMAP) Amplitude from extensor digitorum brevis (EDB) with the reference electrode in the standard location at the base of the ipsilateral 5th toe after injection of BoNT/A into EDB compared with before injection of BoNT/A. Each CMAP represents the mean of 3 individual measurements of the CMAP at that timepoint. In order to facilitate comparison from one subject to the next, the CMAP is then converted into percent change from baseline for that subject. CMAP percent change is then correlated with the percent change in the Surface Electromyography as measured by the Mean Rectified Voltage with 200 millisecond window at the same time points after injection. Group with injection of 20 units BoNT/A is used.
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: percent change from baseline
Groups:
- Surface EMG MRV-200 With Botulinum Toxin Type A, 20 Units: Surface Electromyography (Surface EMG) measured as the MRV (Mean Rectified Voltage) with 200 ms interval
  Single intramuscular (into extensor digitorum brevis muscle of the foot) dose of Botulinum toxin type A, 20 units
  Botulinum Toxin, Type A: 20 units, single dose, intramuscular in right EDB muscle
Arm/Group | CMAP (Standard) With Botulinum Toxin Type A, 20 Units | Surface EMG MRV-200 With Botulinum Toxin Type A, 20 Units
Number analyzed (Participants) | 5 | 5
percent change from baseline
  Day 4 | -53.81 (21.81) | -37.35 (21.98)
  Day 14 | -63.78 (21.77) | -49.49 (28.49)
  Month 4 | -48.38 (26.16) | -38.44 (9.32)
Statistical Analysis 1: Comparison: CMAP (Standard) With Botulinum Toxin Type A, 20 Units vs Surface EMG MRV-200 With Botulinum Toxin Type A, 20 Units; Day 4; Test type: Superiority or Other; p = 0.0374, Spearman Correlation Test; r value = 0.9
Statistical Analysis 2: Comparison: CMAP (Standard) With Botulinum Toxin Type A, 20 Units vs Surface EMG MRV-200 With Botulinum Toxin Type A, 20 Units; Day 14; Test type: Superiority or Other; p = 0.188, Spearman Correlation Test; r value = 0.7
Statistical Analysis 3: Comparison: CMAP (Standard) With Botulinum Toxin Type A, 20 Units vs Surface EMG MRV-200 With Botulinum Toxin Type A, 20 Units; Month 4; Test type: Superiority or Other; p = 0.505, Spearman Correlation Test; r value = 0.4

12. Secondary Outcome: Correlation in Percent Change of the CMAP (With "Inactive" Reference Electrode Location) From EDB After vs. Before Botulinum Toxin Injection Into EDB vs. Percent Change Surface Electromyography (as Measured by Root Mean Squared With 1000 ms Window).
Description: Measure the percent change of the Compound Muscle Action Potential (CMAP) Amplitude from extensor digitorum brevis (EDB) with the reference electrode in an "inactive" location at the ipsilateral medial malleolus after injection of BoNT/A into EDB compared with before injection of BoNT/A. Each CMAP represents the mean of 3 individual measurements of the CMAP at that timepoint. In order to facilitate comparison from one subject to the next, the CMAP is then converted into percent change from baseline for that subject. CMAP percent change is then correlated with the percent change in the Surface Electromyography as measured by the Root Mean Squared with 1000 millisecond window at the same time points after injection. Group with injection of 20 units BoNT/A is used.
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: percent change from baseline
Groups:
- CMAP ("Inactive") With Botulinum Toxin Type A, 20 Units: Compound muscle action potential (CMAP) with reference electrode in an "inactive" location at the ipsilateral medial malleolus
  Single intramuscular (into extensor digitorum brevis muscle of the foot) dose of Botulinum toxin type A, 20 units
  Botulinum Toxin, Type A: 20 units, single dose, intramuscular in right EDB muscle
Arm/Group | CMAP ("Inactive") With Botulinum Toxin Type A, 20 Units | Surface EMG RMS-1000 With Botulinum Toxin Type A, 20 Units
Number analyzed (Participants) | 5 | 5
percent change from baseline
  Day 4 | -67.37 (29.18) | -42.43 (19.82)
  Day 14 | -74.00 (24.46) | -52.35 (27.17)
  Month 4 | -52.40 (33.13) | -39.76 (11.26)
Statistical Analysis 1: Comparison: CMAP ("Inactive") With Botulinum Toxin Type A, 20 Units vs Surface EMG RMS-1000 With Botulinum Toxin Type A, 20 Units; Day 4; Test type: Superiority or Other; p < 0.0001, Spearman Correlation Test; r value = 0.99
Statistical Analysis 2: Comparison: CMAP ("Inactive") With Botulinum Toxin Type A, 20 Units vs Surface EMG RMS-1000 With Botulinum Toxin Type A, 20 Units; Day 14; Test type: Superiority or Other; p = 0.0374, Spearman Correlation Test; r value = 0.9
Statistical Analysis 3: Comparison: CMAP ("Inactive") With Botulinum Toxin Type A, 20 Units vs Surface EMG RMS-1000 With Botulinum Toxin Type A, 20 Units; Month 4; Test type: Superiority or Other; p = 0.104, Spearman Correlation Test; r value = 0.8

13. Secondary Outcome: Correlation in Percent Change of the CMAP (With "Inactive" Reference Electrode Location) From EDB After vs. Before Botulinum Toxin Injection Into EDB vs. Percent Change Surface Electromyography (as Measured by Root Mean Squared With 500 ms Window).
Description: Measure the percent change of the Compound Muscle Action Potential (CMAP) Amplitude from extensor digitorum brevis (EDB) with the reference electrode in an "inactive" location at the ipsilateral medial malleolus after injection of BoNT/A into EDB compared with before injection of BoNT/A. Each CMAP represents the mean of 3 individual measurements of the CMAP at that timepoint. In order to facilitate comparison from one subject to the next, the CMAP is then converted into percent change from baseline for that subject. CMAP percent change is then correlated with the percent change in the Surface Electromyography as measured by the Root Mean Squared with 500 millisecond window at the same time points after injection. Group with injection of 20 units BoNT/A is used.
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: percent change from baseline
Arm/Group | CMAP ("Inactive") With Botulinum Toxin Type A, 20 Units | Surface EMG RMS-500 With Botulinum Toxin Type A, 20 Units
Number analyzed (Participants) | 5 | 5
percent change from baseline
  Day 4 | -67.37 (29.18) | -42.09 (21.19)
  Day 14 | -74.00 (24.46) | -51.94 (28.01)
  Month 4 | -52.40 (33.13) | -40.67 (11.48)
Statistical Analysis 1: Comparison: CMAP ("Inactive") With Botulinum Toxin Type A, 20 Units vs Surface EMG RMS-500 With Botulinum Toxin Type A, 20 Units; Day 4; Test type: Superiority or Other; p < 0.0001, Spearman Correlation Test; r value = 0.99
Statistical Analysis 2: Comparison: CMAP ("Inactive") With Botulinum Toxin Type A, 20 Units vs Surface EMG RMS-500 With Botulinum Toxin Type A, 20 Units; Day 14; Test type: Superiority or Other; p = 0.0374, Spearman Correlation Test; r value = 0.9
Statistical Analysis 3: Comparison: CMAP ("Inactive") With Botulinum Toxin Type A, 20 Units vs Surface EMG RMS-500 With Botulinum Toxin Type A, 20 Units; Month 4; Test type: Superiority or Other; p = 0.0374, Spearman Correlation Test; r value = 0.9

14. Secondary Outcome: Correlation in Percent Change of the CMAP (With "Inactive" Reference Electrode Location) From EDB After vs. Before Botulinum Toxin Injection Into EDB vs. Percent Change Surface Electromyography (as Measured by Root Mean Squared With 200 ms Window).
Description: Measure the percent change of the Compound Muscle Action Potential (CMAP) Amplitude from extensor digitorum brevis (EDB) with the reference electrode in an "inactive" location at the ipsilateral medial malleolus after injection of BoNT/A into EDB compared with before injection of BoNT/A. Each CMAP represents the mean of 3 individual measurements of the CMAP at that timepoint. In order to facilitate comparison from one subject to the next, the CMAP is then converted into percent change from baseline for that subject. CMAP percent change is then correlated with the percent change in the Surface Electromyography as measured by the Root Mean Squared with 200 millisecond window at the same time points after injection. Group with injection of 20 units BoNT/A is used.
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: percent change from baseline
Arm/Group | CMAP ("Inactive") With Botulinum Toxin Type A, 20 Units | Surface EMG RMS-200 With Botulinum Toxin Type A, 20 Units
Number analyzed (Participants) | 5 | 5
percent change from baseline
  Day 4 | -67.37 (29.18) | -39.89 (22.65)
  Day 14 | -74.00 (24.46) | -51.75 (28.52)
  Month 4 | -52.40 (33.13) | -39.90 (12.43)
Statistical Analysis 1: Comparison: CMAP ("Inactive") With Botulinum Toxin Type A, 20 Units vs Surface EMG RMS-200 With Botulinum Toxin Type A, 20 Units; Day 4; Test type: Superiority or Other; p < 0.0001, Spearman Correlation Test; r value = 0.99
Statistical Analysis 2: Comparison: CMAP ("Inactive") With Botulinum Toxin Type A, 20 Units vs Surface EMG RMS-200 With Botulinum Toxin Type A, 20 Units; Day 14; Test type: Superiority or Other; p = 0.0374, Spearman Correlation Test; r value = 0.9
Statistical Analysis 3: Comparison: CMAP ("Inactive") With Botulinum Toxin Type A, 20 Units vs Surface EMG RMS-200 With Botulinum Toxin Type A, 20 Units; Month 4; Test type: Superiority or Other; p = 0.188, Spearman Correlation Test; r value = 0.7

15. Secondary Outcome: Correlation in Percent Change of the CMAP (With "Inactive" Reference Electrode Location) From EDB After vs. Before Botulinum Toxin Injection Into EDB vs. Percent Change Surface Electromyography (as Measured by Mean Rectified Voltage With 1000 ms Window).
Description: Measure the percent change of the Compound Muscle Action Potential (CMAP) Amplitude from extensor digitorum brevis (EDB) with the reference electrode in an "inactive" location at the ipsilateral medial malleolus after injection of BoNT/A into EDB compared with before injection of BoNT/A. Each CMAP represents the mean of 3 individual measurements of the CMAP at that timepoint. In order to facilitate comparison from one subject to the next, the CMAP is then converted into percent change from baseline for that subject. CMAP percent change is then correlated with the percent change in the Surface Electromyography as measured by the Mean Rectified Voltage with 1000 millisecond window at the same time points after injection. Group with injection of 20 units BoNT/A is used.
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: percent change from baseline
Arm/Group | CMAP ("Inactive") With Botulinum Toxin Type A, 20 Units | Surface EMG MRV-1000 With Botulinum Toxin Type A, 20 Units
Number analyzed (Participants) | 5 | 5
percent change from baseline
  Day 4 | -67.37 (29.18) | -40.92 (18.90)
  Day 14 | -74.00 (24.46) | -51.03 (26.56)
  Month 4 | -52.40 (33.13) | -37.86 (9.45)
Statistical Analysis 1: Comparison: CMAP ("Inactive") With Botulinum Toxin Type A, 20 Units vs Surface EMG MRV-1000 With Botulinum Toxin Type A, 20 Units; Day 4; Test type: Superiority or Other; p < 0.0001, Spearman Correlation Test; r value = 0.99
Statistical Analysis 2: Comparison: CMAP ("Inactive") With Botulinum Toxin Type A, 20 Units vs Surface EMG MRV-1000 With Botulinum Toxin Type A, 20 Units; Day 14; Test type: Superiority or Other; p = 0.0374, Spearman Correlation Test; r value = 0.9
Statistical Analysis 3: Comparison: CMAP ("Inactive") With Botulinum Toxin Type A, 20 Units vs Surface EMG MRV-1000 With Botulinum Toxin Type A, 20 Units; Month 4; Test type: Superiority or Other; p = 0.391, Spearman Correlation Test; r value = 0.5

16. Secondary Outcome: Correlation in Percent Change of the CMAP (With "Inactive" Reference Electrode Location) From EDB After vs. Before Botulinum Toxin Injection Into EDB vs. Percent Change Surface Electromyography (as Measured by Mean Rectified Voltage With 500 ms Window).
Description: Measure the percent change of the Compound Muscle Action Potential (CMAP) Amplitude from extensor digitorum brevis (EDB) with the reference electrode in an "inactive" location at the ipsilateral medial malleolus after injection of BoNT/A into EDB compared with before injection of BoNT/A. Each CMAP represents the mean of 3 individual measurements of the CMAP at that timepoint. In order to facilitate comparison from one subject to the next, the CMAP is then converted into percent change from baseline for that subject. CMAP percent change is then correlated with the percent change in the Surface Electromyography as measured by the Mean Rectified Voltage with 500 millisecond window at the same time points after injection. Group with injection of 20 units BoNT/A is used.
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: percent change from baseline
Arm/Group | CMAP ("Inactive") With Botulinum Toxin Type A, 20 Units | Surface EMG MRV-500 With Botulinum Toxin Type A, 20 Units
Number analyzed (Participants) | 5 | 5
percent change from baseline
  Day 4 | -67.37 (29.18) | -40.44 (20.00)
  Day 14 | -74.00 (24.46) | -50.72 (27.40)
  Month 4 | -52.40 (33.13) | -39.22 (9.42)
Statistical Analysis 1: Comparison: CMAP ("Inactive") With Botulinum Toxin Type A, 20 Units vs Surface EMG MRV-500 With Botulinum Toxin Type A, 20 Units; Day 4; Test type: Superiority or Other; p < 0.0001, Spearman Correlation Test; r value = 0.99
Statistical Analysis 2: Comparison: CMAP ("Inactive") With Botulinum Toxin Type A, 20 Units vs Surface EMG MRV-500 With Botulinum Toxin Type A, 20 Units; Day 14; Test type: Superiority or Other; p = 0.0374, Spearman Correlation Test; r value = 0.9
Statistical Analysis 3: Comparison: CMAP ("Inactive") With Botulinum Toxin Type A, 20 Units vs Surface EMG MRV-500 With Botulinum Toxin Type A, 20 Units; Month 4; Test type: Superiority or Other; p = 0.0374, Spearman Correlation Test; r value = 0.9

17. Secondary Outcome: Correlation in Percent Change of the CMAP (With "Inactive" Reference Electrode Location) From EDB After vs. Before Botulinum Toxin Injection Into EDB vs. Percent Change Surface Electromyography (as Measured by Mean Rectified Voltage With 200 ms Window).
Description: Measure the percent change of the Compound Muscle Action Potential (CMAP) Amplitude from extensor digitorum brevis (EDB) with the reference electrode in an "inactive" location at the ipsilateral medial malleolus after injection of BoNT/A into EDB compared with before injection of BoNT/A. Each CMAP represents the mean of 3 individual measurements of the CMAP at that timepoint. In order to facilitate comparison from one subject to the next, the CMAP is then converted into percent change from baseline for that subject. CMAP percent change is then correlated with the percent change in the Surface Electromyography as measured by the Mean Rectified Voltage with 200 millisecond window at the same time points after injection. Group with injection of 20 units BoNT/A is used.
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: percent change from baseline
Arm/Group | CMAP ("Inactive") With Botulinum Toxin Type A, 20 Units | Surface EMG MRV-200 With Botulinum Toxin Type A, 20 Units
Number analyzed (Participants) | 5 | 5
percent change from baseline
  Day 4 | 67.37 (29.18) | -37.35 (21.98)
  Day 14 | -74.00 (24.46) | -49.49 (28.49)
  Month 4 | -52.40 (33.13) | -38.44 (9.32)
Statistical Analysis 1: Comparison: CMAP ("Inactive") With Botulinum Toxin Type A, 20 Units vs Surface EMG MRV-200 With Botulinum Toxin Type A, 20 Units; Day 4; Test type: Superiority or Other; p < 0.0001, Spearman Correlation Test; r value = 0.99
Statistical Analysis 2: Comparison: CMAP ("Inactive") With Botulinum Toxin Type A, 20 Units vs Surface EMG MRV-200 With Botulinum Toxin Type A, 20 Units; Day 14; Test type: Superiority or Other; p = 0.0374, Spearman Correlation Test; r value = 0.9
Statistical Analysis 3: Comparison: CMAP ("Inactive") With Botulinum Toxin Type A, 20 Units vs Surface EMG MRV-200 With Botulinum Toxin Type A, 20 Units; Month 4; Test type: Superiority or Other; p = 0.505, Spearman Correlation Test; r value = 0.4

ADVERSE EVENTS:
Arm/Group | Botulinum Toxin Type A, 20 Units | Botulinum Toxin, Type A, 2 Units | Placebo
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/4 | 0/4
Other Adverse Events (participants affected / at risk) | 3/5 | 1/4 | 0/4
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Botulinum Toxin Type A, 20 Units (N=5) | Botulinum Toxin, Type A, 2 Units (N=4) | Placebo (N=4)
Decreased sensation (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Flu like symptoms (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 0 (0)
Mild Headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes